CLINICAL TRIAL: NCT02579148
Title: Collagen Scaffolds Loaded With Human Umbilical Cord Mesenchymal Stem Cells for the Improvement of Erectile Function in Men With Diabetes
Brief Title: Collagen Scaffolds Loaded With HUCMSCs for the Improvement of Erectile Function in Men With Diabetes
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Leilei Zhu (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor-Investigator, Leilei Zhu, science and technology department head, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DTH-922-DYT
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2015-10

CONDITIONS: Erectile Dysfunction; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: erectile dysfunction; stem cell; collagen scaffold
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- HUCMSC injection (Experimental): once intracavernous injection of 15,000,000 Human Umbilical Cord Mesenchymal Stem Cells
  Interventions: Biological: HUCMSC injection
- collagen scaffolds/HUCMSC injection (Experimental): once intracavernous injection of collagen scaffolds loaded with 15,000,000 Human Umbilical Cord Mesenchymal Stem Cells
  Interventions: Biological: collagen scaffolds/HUCMSC injection

INTERVENTIONS:
Biological: HUCMSC injection — The subjects will receive intracavernous injection of HUCMSC.'
  Arms: HUCMSC injection
Biological: collagen scaffolds/HUCMSC injection — The subjects will receive intracavernous injection of the mixture of collagen scaffolds and HUCMSC respectively.'
  Arms: collagen scaffolds/HUCMSC injection

SUMMARY:
The intent of this clinical study is to answer the questions: 1) is the proposed treatment feasible; 2) is treatment effective in improving the disease pathology of patients with diagnosed diabetic erectile dysfunction.

DETAILED DESCRIPTION:
Intracavernous transplantation of stem cells has been shown to improve erectile function in some preclinical studies. However, inadequate cell homing to damaged sites limited its functions. The investigators explore the effect of HUCMSC on improving erectile function of diabetic men, and whether collagen scaffolds contribute to long-term cell retention in the corpus cavernous and improves erectile function of diabetic men.

ELIGIBILITY:
Inclusion Criteria:

1. type 1 or 2 diabetes,blood glucose controlled well, no effective with oral PDE-5i;
2. have a consistent partner who is willing to engage in sexual activity more than twice per month during the study;
3. males age 20-65 years;
4. IIEF-5 score is under 16;
5. penile arterial insufficiency or venous leakage (doppler): PSV <25 cm/sec, or PSV >25 cm/sec, EDV>5cm/sec, RI<0, 75;
6. HbA1c is between 6.5% 10%;
7. physical examination with no abnormalities;
8. who is willing to consent to participate in the study follow-up;
9. willing to limit alcohol intake eliminate use of recreational drugs for sexual encounters.

Exclusion Criteria:

1. severe cardiovascular disease(angina, arrhythmia, cardiac failure, stroke), kidney failure, respiratory failure; history of malignancy;
2. positive for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) syphilis test;
3. Testosterone level is less than 200ng/dl;
4. serum AST/ALT >3*upper limit of normal or creatinine >1.5*upper limit of normal;
5. HbA1c exhibit greater than 10%;
6. in the investigators judgment, with clinical significance of penis abnormalities, or has received penile prosthesis implantation surgery;
7. patients partner is trying to conceive during the trial period;
8. exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study;
9. unwilling and/or not able to give written informed consent.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Improvements in IIEF scores | 1,3,6,9 and 12 months
  The subjects must fill in the questionnaire of IIEF-5 every visit to evaluate erectile function.

SECONDARY OUTCOMES:
Penile colour Doppler ultrasonography combined with prostaglandin-E1 injection | 1,3,6,9 and 12 months
Safety and Tolerability assessed by Adverse Events | 1 month after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- Drum Tower Hospital, Nanjing, Jiangsu, China